CLINICAL TRIAL: NCT01871259
Title: Clinical Predictors of Apnea-hypopnea During Propofol Sedation in Patients Undergoing Spinal Anaesthesia
Brief Title: Clinical Predictors of Apnea-hypopnea During Propofol Sedation
Acronym: sleeposa
Status: Terminated | Type: Observational
Why Stopped: Finished
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Jin Lee, professor, Samsung Medical Center
Other Study IDs: sleeposa
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Sleep Apnea
Keywords: Sedation, sleep apnea, propofol
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To relate two different predictive values of sleep apnea: the STOP score (snoring while sleeping, daytime tiredness, observed breathing stoppages, and high blood pressure) and the estimated respiratory disturbance index (eRDI) with the occurrence of apnea-hypopnea during propofol sedation,thirty four middle-aged male patients who underwent urologic surgery under spinal anaesthesia will be enrolled. Before surgery, patients will be asked to complete a STOP-questionnaire. The eRDI will be calculated using the modified Mallampati's grade, tonsil grade, and the body mass index. After performing spinal anaesthesia, propofol will be infused and adjusted to BIS 70-75. An ApneaLinkTM, which measures airflow through a nasal cannula, will be then applied to estimate the level of apnea-hypopnea.

DETAILED DESCRIPTION:
The investigators will evaluate correlation between STOP scor and AHI(apnea hypopnea index) or eRDI and AHI. After then the investigators will compare AHI severity between high risk group and low risk group subgrouped according to STOP score or eRDI.

ELIGIBILITY:
Inclusion Criteria:

* Thirty four males who underwent spinal anaesthesia for transurethral resection of the bladder (TURB) or prostate (TURP) were enrolled in this studyInclusion criteria were American Society of Anaesthesiologists (ASA) physical status of 1-2, and ages of more than 40 years.

Exclusion Criteria:

* Patients with electrocardiographic or simple chest radiographic abnormalities or who had taken medication that could affect their sleep patterns were excluded.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We expected a correlation coefficient of ~0.5 in this study, which meant that for a level of significance of 5% and a power of 80%, we required 29 analyzable subjects. Based on a predicted exclusion rate of 15%, 34 patients were included.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index | 1hour
  After surgery, an ApneaLinkTM was connected to a personal computer to record and auto-analyze AHIs. Aopnea was defined as a cessation of airflow for 10s or longer. Hypopnea was defined as a greater than 50% reduction in airflow for 10s or longer. AHI was defined as the number of aopnea and hypopnea incidents per hour.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Jin Lee, Professor, Principal Investigator — : Department of Anaesthesiology and Pain Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine